CLINICAL TRIAL: NCT02160041
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 6 - BGJ398 for Patients With Tumors With FGFR Genetic Alterations
Brief Title: BGJ398 for Patients With Tumors With FGFR Genetic Alterations
Acronym: CBGJ398XUS04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398XUS04
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor; Hematologic Malignancies
Keywords: Solid tumor malignancy; hematologic malignancy; mutation; translocations; amplifications,; fusions; signature; FGFR; ligand; BGJ398
MeSH Terms: conditions — Hematologic Neoplasms | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BGJ398 (Experimental): BGJ398 was dosed on a flat scale of 125 mg (e.g., 1 x 100 mg and 1 x 25 mg capsules) once daily for the first 21 days of the 28-day cycle (3 weeks on, 1 week off in a cycle). A complete treatment cycle is defined as 28 days.
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398 — BGJ398 was dosed on a flat scale of 125 mg (e.g., 1 x 100 mg and 1 x 25 mg capsules) once daily for the first 21 days of the 28-day cycle (3 weeks on, 1 week off in a cycle). A complete treatment cycle is defined as 28 days.

SUMMARY:
The purpose of this signal seeking study was to determine whether treatment with BGJ398 demonstrates sufficient efficacy in select FGFR pathway-regulated solid tumors and/or hematologic malignancies to warrant further study.

ELIGIBILITY:
Inclusion Criteria:

Patient has a confirmed diagnosis of a select solid tumor (except with a primary diagnosis of Urothelial cell carcinoma, Cholangiocarcinoma, Endometrial cancer, and Glioblastoma multiforme) or hematologic malignancies and is in need of treatment because of progression or relapse.

Patient's tumor has been evaluated and pre-identified as having a tumor with a FGFR genetic alteration. The qualifying alteration must be assessed and reported by a CLIA-certified laboratory.

Patient must have received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options are anticipated to result in a durable remission.

Patient must have progressive and measurable disease per RECIST 1.1. or other appropriate hematological response criteria.

Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

Patient has received prior treatment with BGJ398

Patients with Central Nervous System (CNS) metastasis or leptomeningeal carcinomatosis

Patient has received chemotherapy or other anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug.

Patients with acute or chronic pancreatitis

Patients with impaired cardiac function or clinically significant cardiac diseases

History and/or current evidence of extensive tissue calcification

Use of medications that increase serum levels of phosphorus and/or calcium

Current evidence of corneal or retinal disorder/keratopathy

History and/or current evidence of renal or endocrine alterations of calcium/phosphate homeostasis

Patients with another primary malignancy within 3 years prior to starting study treatment, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Alabama Oncology St. Vincent's Birmingham, Birmingham, Alabama
  - North County Oncology Medical Clinic Inc, Oceanside, California
  - San Francisco General Hospital San Francisco Gen Hosp (7), San Francisco, California
  - Rocky Mountain Cancer Centers Rocky Mountain Cancer Ctr (50), Greenwood Village, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Florida Cancer Specialists Florida Cancer Specialists 36, Fort Myers, Florida
  - University of Miami Sylvester Comprehensive Cancer, Miami, Florida
  - NorthWest Georgia Oncology Centers NW Georgia Oncology, Marietta, Georgia
  - Harbin Clinic Medical Oncology Clin. Res., Rome, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Indiana University Indiana Univ. - Purdue Univ., Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium No. Indiana Cancer Res., South Bend, Indiana
  - University of Louisville / James Graham Brown Cancer Center SC, Louisville, Kentucky
  - St. Agnes Hospital St. Agnes Hospital (2), Baltimore, Maryland
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Cancer and Hematology Centers of West Michigan Dept. of Oncology, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, P.A. Minnesota Oncology Hem (27), Minneapolis, Minnesota
  - Research Medical Center Research Med Center (2), Kansas City, Missouri
  - Billings Clinic Billings Clinic (8), Billings, Montana
  - Dartmouth Hitchcock Medical Center Dartmouth Hitchcock - Lebanon, Bedford, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Waverly Hematology Oncology, Cary, North Carolina
  - University of N C at Chapel Hill Physician Office Building, Chapel Hill, North Carolina
  - Duke University Medical Center Seeley G. Mudd Bldg., Durham, North Carolina
  - Wake Forest Baptist Health Hem & Onc Medical Center, Winston-Salem, North Carolina
  - Sanford Hematology Oncology, Fargo, North Dakota
  - Oncology Hematology Care Inc Oncology Hematology Care 2, Cincinnati, Ohio
  - University Hospitals of Cleveland Seidman Cancer Center University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio
  - Bend Memorial Clinic Bend Mem. Clinic, Bend, Oregon
  - Northwest Cancer Specialists Northwest Cancer, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Cancer Treatment Centers of America Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute Hillman Cancer Center (2), Pittsburgh, Pennsylvania
  - Rhode Island Hospital Rhode Island Hosp. (2), Providence, Rhode Island
  - Sanford University of South Dakota Medical Center Sanford Health, Sioux Falls, South Dakota
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - Tennessee Oncology Tennessee Oncology (3), Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Oncology Consultants Oncology Group, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Texas Oncology, McAllen, Texas
  - Cancer Therapy & Research Center UT Health Science Center Oncology Dept., San Antonio, Texas
  - Texas Oncology Cancer Care & Research Center Texas Oncology, Waco, Texas
  - Deke Slayton Cancer Center Deke Slayton Cancer Center (2), Webster, Texas
  - Intermountain Medical Center Intermountain Healthcare, Murray, Utah
  - Northern Utah Cancer Associates Northern Utah Assoc (3), Ogden, Utah
  - University of Utah / Huntsman Cancer Institute SC-2, Salt Lake City, Utah
  - Utah Cancer Specialists Utah Cancer Specialists (11), Salt Lake City, Utah
  - Virginia Cancer Specialists Fairfax Northern Virginia, Fairfax, Virginia
  - Shenandoah Oncology Shenandoah Oncology (5), Winchester, Virginia
  - Northwest Medical Specialties NW Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BGJ398
Started | 84
Completed | 0
Not Completed | 84
Not completed — Adverse Event | 11
Not completed — Death | 2
Not completed — disease progression | 57
Not completed — Protocol Violation | 1
Not completed — non-compliance with study | 1
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 8
Not completed — study terminated by by sponsor | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS included all enrolled patients who received at least 1 dose of study drug. The FAS was the primary set for efficacy analyses.
Arm/Group | BGJ398
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12.08)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 54
  >=65-<75 years | 21
  >=75 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 74
  Black | 6
  Asian | 1
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) Associated With BGJ398 Treatment
Description: Tumor Response: Overall response rate (ORR) and clinical benefit rate (CBR) for solid tumor (non-lymphoma) which excludes 3 TIO and 1 Lymphoma patients (hence 80 patients and not 84)
  Clinical benefit rate for patients with solid tumors were assessed using RECIST 1.1 and include responses of CR or PR or SD. For hematologic tumors other appropriate hematological response criteria may apply
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 16 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BGJ398
Number analyzed (Participants) | 80
Participants
  Complete response (CR) | 0
  Partial response (PR) | 6
  Progressive disease (PD) | 54
  Stable disease (SD) | 7
  Non-evaluable (NE) | 13
  Overall response rate (ORR: CR + PR) | 6
  Clinical benefit rate (CBR: CR+PR+SD) | 12

2. Secondary Outcome: Overall Response (OR) or Partial Response (PR) or Greater
Description: The key secondary endpoint, OR, was determined by Investigator assessment for each tumor assessment and defined as responses of CR and PR per RECIST version 1.1.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: baseline and every 8 weeks until disease progression or end of treatment, assessed up to 24 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | BGJ398
Number analyzed (Participants) | 84
participants | 6 [2.8 to 15.6]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Kaplan-Meier estimates of PFS timing, months
  Progression free survival (PFS) is defined as the time from the date of first dose to the date of first documented disease progression or relapse or death due to any cause
Time Frame: every 8 weeks until death, assessed up to 24 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGJ398
Number analyzed (Participants) | 82
months | 1.8 [1.8 to 2.0]

4. Secondary Outcome: Kaplan-Meier Estimates of PFS Rate, % (95% CI)
Time Frame: Months 1, 2, 3, 4, 5, 6, 12, 18, 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | BGJ398
Number analyzed (Participants) | 82
percent of participants
  Month 1 | 88.0 [78.2 to 93.6]
  Month 2 | 38.0 [27.0 to 48.9]
  Month 3 | 32.3 [21.9 to 43.0]
  Month 4 | 20.0 [11.5 to 30.1]
  Month 5 | 15.4 [8.0 to 24.9]
  Month 6 | 12.3 [5.8 to 21.3]
  Month 12 | 10.2 [4.3 to 19.2]
  Month 18 | 6.1 [1.8 to 14.5]
  Month 24 | 0.0 [0.0 to 0.0]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause
Time Frame: every 8 weeks until death, assessed up to 36 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BGJ398
Number analyzed (Participants) | 84
months | 6.2 [4.4 to 9.8]

6. Secondary Outcome: Kaplan-Meier Estimates of Survival Rate, % (95% CI)
Description: Overall survival (OS) is the time from the date of start of treatment to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last contact.
Time Frame: months 3, 6, 9, 12, 24
Population: FAS
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | BGJ398
Number analyzed (Participants) | 84
percent of participants
  Month 3 | 75.9 [64.9 to 83.9]
  Month 6 | 50.1 [38.6 to 60.6]
  Month 9 | 39.4 [28.5 to 50.1]
  Month 12 | 35.1 [24.6 to 45.8]
  Month 24 | 19.5 [10.5 to 30.5]

7. Secondary Outcome: Number of Participants With 99 Day Minimum Duration of Response (DOR)
Description: The duration of response (PR or greater) applies only to patients whose best response was PR or greater. It is defined as the Ttime from the first documented response to the date first documented disease progression or relapse or death due to any cause
Time Frame: baseline and every 8 weeks until disease progression or end of treatment, assessed up to 24 months
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | BGJ398
Number analyzed (Participants) | 84
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to maximum of 26.6 months
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 26.6 months
Arm/Group | BGJ398
All-Cause Mortality (participants affected / at risk) | 11/83
Serious Adverse Events (participants affected / at risk) | 33/83
Other Adverse Events (participants affected / at risk) | 81/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BGJ398 (N=83)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Enterovesical fistula (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Blood creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Coma (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BGJ398 (N=83)
Anaemia (Blood and lymphatic system disorders) | 9
Dry eye (Eye disorders) | 16
Punctate keratitis (Eye disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 26
Diarrhoea (Gastrointestinal disorders) | 20
Dry mouth (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 6
Glossodynia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 26
Oral pain (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 5
Fatigue (General disorders) | 44
Mucosal inflammation (General disorders) | 15
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 7
Conjunctivitis (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 12
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 10
Blood alkaline phosphatase increased (Investigations) | 9
Blood creatinine increased (Investigations) | 17
Blood phosphorus increased (Investigations) | 14
Gamma-glutamyltransferase increased (Investigations) | 5
Lipase increased (Investigations) | 5
Weight decreased (Investigations) | 15
Decreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 12
Hypercalcaemia (Metabolism and nutrition disorders) | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 47
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 12
Hyponatraemia (Metabolism and nutrition disorders) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 17
Headache (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 8
Nail discolouration (Skin and subcutaneous tissue disorders) | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 8
Onychomadesis (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02160041/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT02160041/SAP_001.pdf